CLINICAL TRIAL: NCT07239076
Title: Unstimulated Gluteus Maximus Sphincteroplasty for Treatment of Bowel Incontinence
Brief Title: Unstimulated Gluteus Maximus Sphincteroplasty for Treatment of Bowel Incontinnence Case Series Study
Acronym: USGMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelrazak Mohamed Ahmed, Unstimulatedgulteus maximus sphincteroplasty for treatment of bowel incontinence, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anal sphincteroplasty
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Bowel Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Age not below 9 years (Experimental): Surgery target people not below the age of 9 yearsLower gluteal crease incision and lower third fibers taken with neovascular bundle and suturing on contralateral ischial tuberosity to make external sphincter and make neosphincter
  Interventions: Procedure: Unstimulated gluteus maximus sphincteroplasty

INTERVENTIONS:
Procedure: Unstimulated gluteus maximus sphincteroplasty — Surgery done under general anethesia prone jacknige postion .. incsion made along lower gluteal crease to take lower third fibers including neurovascular bundle and dicussating subcutaneusly around anus and suturing on contralateral ischial tuberosity

SUMMARY:
Unstimlated gluteus maximus sphincteroplasty for treatment of bowle incontinence

DETAILED DESCRIPTION:
Surgery to treat patient with bowel incontinence by using unstimulated gluteus maximus muslce in creating neosphincter by dicussating lower third of muscle with neovascular bundle and suturing on contralateral side ischial tuberosity

ELIGIBILITY:
Inclusion Criteria:

* patients with severe fecal incontinence refractory to medical treatment
* loss of native anal sphincter confirmed by MRI
* patients deemed suitable for unstimulated gluteus maximus sphincteroplasty

Exclusion Criteria:

* amyotrophic lateral sclerosis
* severe scarring of bilateral gluteus maximus
* pelvic fracture with injury of internal illiac vessels

Ages: 9 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of fecal incontinence | 6 months
  Improvement of fecal incontince assessed by cleveland clinic florida fecal incontinnence score <7
Improvement of fecal incontinence | 6 months
  Improvement of fecal incontinence assessed by cleveland clinic florida fecal incontinence score at final follow uo <7

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Refaat Shehata, Assistant professor, Principal Investigator — Assiut University
Locations (1):
- Assiut hospital university, Asyut, University, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Treat patients with fecal incontinence
Supporting Information: Study Protocol
Time Frame: Start date 2025 End date 2028
Access Criteria: Everyone
URL: http://Clevelandclinicfloridafecalincontinencsscore.com

REFERENCES:
- [Result] Dexter T, WalshawJ ,Winny H,LeoA
- See also: Treatment of bowel incontinence — https://pmc.ncbi.nlm.nih.gov/articles/PMC10049812/
- See also: Treatment of fecal incontinence — https://pmc.ncbi.nlm.nih.gov/articles/PMC10049812/
- Available data/document: Informed Consent Form: AssitU — https://pmc.ncbi.nlm.nih.gov/articles/PMC10049812/ — For treatment